CLINICAL TRIAL: NCT00147433
Title: Are IQs Low in Offspring of Euthyroid Women With Low T4?
Brief Title: The Effect of Thyroid Hormone Levels in Pregnant Women on the Intelligence Quotient (IQ) of Their Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: R01HD044111 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2006-03-31 (Estimated); Status verified 2005-09

CONDITIONS: Child Development Disorders; Pregnancy; Subclinical Hypothyroidism
Keywords: free thyroxine; pregnancy; fetal brain development; thyroid stimulating hormone; IQ
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
This study is designed to test the hypothesis that the level of the thyroid hormone thyroxine (specifically, free thyroxine, FT4) circulating in the blood of pregnant women is the key thyroid-related factor to influence early fetal brain development. The investigators will recruit 5000 pregnant women with clinically normal thyroid function (normal thyroid stimulating hormone levels) in the second trimester. After the baby has been born, the investigators will measure FT4 in the second trimester maternal blood sample to identify 100 cases (very low FT4 levels) and 100 matched controls (normal FT4 levels). The children of cases and controls will undergo neurodevelopmental testing at 2 years of age to determine whether IQ differs according to maternal FT4 levels during pregnancy. The potential impact of the study is that if such an effect is found, it might be possible to avoid these adverse developmental consequences in children by designing and testing strategies to identify and treat high risk women.

DETAILED DESCRIPTION:
Summary:

The purpose of the proposed study is to test the hypothesis that the key thyroid-related factor in early fetal brain development is T4 derived from the maternal circulation. According to this hypothesis, low circulating maternal levels of free T4 may adversely influence fetal brain development, even when the mother is clinically euthyroid (i.e. has normal TSH levels).

Specific Aims:

The proposed project aims to determine whether free T4 levels at or below the 3rd centile in euthyroid women during early pregnancy are associated with reduced neuropsychological development in their offspring. We will recruit a cohort of 5,000 pregnant women whose serum samples have been submitted for routine prenatal screening for Down syndrome and neural tube defects in the early second trimester of pregnancy. After the women provide consent, thyroid-stimulating hormone (TSH) measurements will be performed. The women defined as euthyroid by TSH measurement will comprise the study group. Free T4 measurements will be performed on their stored sera after delivery. Then, a nested case-control study design will be used. Inclusion criteria will include: liveborn, singleton infant delivered in Maine at 36 weeks or later, weighing at least 2,500 grams, and with no reported congenital anomalies. Multiple gestations will be excluded. Eligible women with free T4 measurements below the 3rd percentile (cases) will each be matched with a woman/infant pair with normal free T4 measurements (controls). Overall, 100 offspring in each category will undergo neurodevelopmental testing at age 2 years, using a test battery that will focus on language development and attainment of milestones and motor development. The study will have an 80% power to detect a 6 point difference in full scale IQ.

Study Timeline:

Phase 1. Preparation for Recruitment (months 1-4):

Validate reference ranges for TSH and Free T4 Assays; Implement clinical reporting and management system for TSH measurements; design and implement a Data Management System; develop Provider and patient materials; visit offices to introduce the project; develop informed consent.

Phase 2. Active Recruitment (months 4-24):

Recruit 5,000 pregnant women, classified as euthyroid based on second trimester TSH measurements; measure free T4 measured in stored serum aliquots after the pregnancies have delivered.

Phase 3. Identification of Study Subjects (months 18-36):

Identify 100 cases (euthyroid women fulfilling all inclusion criteria and with free T4 measurements at or below the 3rd centile) and 100 matched controls (normal free T4) among the 5,000 euthyroid recruits.

Phase 4. Locate/Recruit Cases and Controls (months 20-38):

Locate and re-recruit the women/infant pairs identified in phase 3; obtain newborn hypothyroidism screening results.

Phase 5. Neurodevelopmental Testing (months 36-58):

Perform neurodevelopmental testing and measure other thyroid analytes (total T4, T3 and thyroid antibodies) in the cases and controls.

Phase 6. Data Analysis (months 59-60):

Compare demographic data, along with pregnancy- and delivery-related information, between case and control mother/child pairs to verify matching and to compare non-matched variables between the two groups. Include covariates that differ significantly between cases and controls (and that might be related to neurodevelopment) in a more refined model to determine whether the unadjusted findings are robust.

Significance:

The knowledge gained from this study will expand our understanding of the role that thyroid hormone plays in normal pregnancy. If the hypothesis under study in this proposal proves to be correct, it will define a broader group of pregnancies in which fetal brain development might be suboptimal. The primary benefit to documenting such a problem would be the opportunity to develop strategies for identifying and treating high risk women to avoid the adverse consequences in their children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female
* Normal TSH in second trimester
* Singleton pregnancy
* Term infant weighing 2500g or more
* No congenital abnormalities noted on birth record
* Delivery in Maine at 36 weeks or later

Exclusion Criteria:

* TSH levels outside normal range in second trimester
* Pre-existing hypothyroidism, treated
* More than one fetus
* Premature and/or low birth weight infant
* Congenital abnormalities noted on birth record

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000
Dates: Start 2004-02; Study Completion 2008-11

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Y. Craig, Ph.D., Principal Investigator — Foundation for Blood Research
Locations (1):
- Foundation for Blood Research, Scarborough, Maine, United States

REFERENCES:
- [Background] Haddow JE, Palomaki GE, Allan WC, Williams JR, Knight GJ, Gagnon J, O'Heir CE, Mitchell ML, Hermos RJ, Waisbren SE, Faix JD, Klein RZ. Maternal thyroid deficiency during pregnancy and subsequent neuropsychological development of the child. N Engl J Med. 1999 Aug 19;341(8):549-55. doi: 10.1056/NEJM199908193410801. PMID 10451459
- [Background] Allan WC, Haddow JE, Palomaki GE, Williams JR, Mitchell ML, Hermos RJ, Faix JD, Klein RZ. Maternal thyroid deficiency and pregnancy complications: implications for population screening. J Med Screen. 2000;7(3):127-30. doi: 10.1136/jms.7.3.127. PMID 11126160